CLINICAL TRIAL: NCT01606865
Title: Does Platelet Inhibition Predict Surgery Related Bleeding in Patients Undergoing Non-Cardiac Surgery During Dual Antiplatelet Therapy
Brief Title: Platelet Inhibition and Bleeding in Patients Undergoing Non-Cardiac Surgery
Acronym: BIANCA
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Principal Investigator, Helfried Metzler, MD, Prof., Medical University of Graz
Other Study IDs: BIANCA
Record Dates: First submitted 2012-05-24; First posted 2012-05-28 (Estimated); Last update posted 2014-10-23 (Estimated); Status verified 2014-10

CONDITIONS: Postoperative Bleeding
MeSH Terms: conditions — Postoperative Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- elective and acute non-cardiac surgery

SUMMARY:
The aim of the study is to evaluate if there is an association between platelet inhibition and surgery-related bleeding in patients undergoing non-cardiac surgery during dual antiplatelet therapy.

ELIGIBILITY:
Inclusion Criteria:

* intake of Clopidogrel, Prasugrel, or Ticagrelor within the last 7 days
* spontaneous bleeding or impeding surgery (major vascular surgery, intraperitoneal or intrathoracic surgery, ENT-surgery, orthopedic or trauma surgery, prostatic surgery)

Exclusion Criteria:

* concomitant medication with warfarin
* renal insufficiency needing dialysis
* concomitant therapy with GPIIB/IIIA Antagonists
* expected duration of operation >30min

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients taking Clopidogrel, Prasugrel, or Ticagrelor within at least 7 days
Sampling Method: Probability Sample
Enrollment: 207 (Actual)
Dates: Start 2010-09; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
increased risk of bleeding (according to TIMI definition) | 24hours postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Helfried Metzler, Prof. Dr., Study Chair — Medical University of Graz
Locations (1):
- Department of Anesthesiology and Intensive Care Medicine, Medical University Graz, Graz, Austria